CLINICAL TRIAL: NCT03558789
Title: Metallic Taste Before, During and After Treatment of Head and Neck Cancer : Etiologies and Impact on Quality of Life
Brief Title: Metallic Taste Before, During and After Treatment of Head and Neck Cancer
Acronym: TORCAD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Valence (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH-CHV-01
Record Dates: First submitted 2018-04-26; First posted 2018-06-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2023-12

CONDITIONS: Metallic Taste
MeSH Terms: conditions — Taste Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MT: patients complaining about metallic taste before, during or after treatment of head and neck cancer.
  Interventions: Biological: bovine lactoferrin
- No-MT: patients not complaining about metallic taste before, during or after treatment of head and neck cancer.
  Interventions: Biological: bovine lactoferrin

INTERVENTIONS:
Biological: bovine lactoferrin — mouthwash

SUMMARY:
Metallic taste in head and neck cancer is widely under-estimated in the literature. Its causes are multiple and poorly defined. Though it has a strong impact on the nutritional status.

The main objective of the TORCAD project is to test the hypothesis that intraoral lipoperoxidation is associated to metallic taste onset before, during and after treatment of head and neck cancer (HNC).

The secondary goals are to evaluate the involvement of others physiopathological factors in metallic taste: (i) additional chemical modification in the saliva; (ii) release of inhibition of the facial nerve on the glossopharyngeal nerve; presence of an intraoral electric current; food pleasantness and acceptability; quality of life.

DETAILED DESCRIPTION:
The objectives of this study are to perform tests and questionnaires. All samples will be non-invasive.

Evaluation of metallic taste (MT) occurrence with a specific questionnaire. In a single patient, MT occurrence may vary according to the time of the study.

1. Oral media modifications 1.1- Salivary functions: basal and stimulated salivary flow will be determined. Immediately after collection, both salivary samples will be stored at -80°C. Twice a year frosted samples will be delivered to the Centre des Sciences du Goût et de l'Alimentation in Dijon, France) by a special transporter. Biochemical analyses of saliva will consist of analyses of candidate markers: malondialdehyde, metabolites (uric acid), ions (Mn2+ and Zn2+), enzymatic activities and key proteins involved in the salivary peroxidation (catalase, superoxide dismutase). All the technics are already validated.

   1.2- Quantification of fungiform papillae in dermatoscopy. The objective of the dermatoscope is placed on the tongue and a snapshot of a predefined surface area will be recorded on both sides of the tongue. The density will be estimated according to an automatic method from the snapshots.

   1.3- Trapping of nasal scents To assess the presence of volatile odorous compounds induced by the oral lipoperoxidation, the nasal scents of the patients will be harvested by a Tenax® trap positioned at the exit of nostril. The operation will be performed without any stimulus, after an iron sulphate mouthwash (artificially inducing MT) and after treatment with lactoferrin mouthwash (chelating agent). The traps will be hermetically closed and sent to the Centre des Sciences du gout et de l'Alimentation in Dijon for analysis by gas chromatography/mass spectrometry. These tests will be performed after psychophysical tests not to distort their results.
2. Psychophysical tests. 2.1- Psychophysical tests of taste intensity will be carried out with two aqueous solutions (one neutral, the other sapid) of each taste (salty, sweet, sour, bitter and umami) and iron sulphate. The solutions will moisten 0.5 cm-diameter filter paper discs that will be deposited on the tongue. For each taste, patients will have to indicate the disc with the strongest and least strong taste. Four locations on the tongue will be tested: one for the territory of the facial nerve (anterior tongue), one for the glossopharyngeal nerve (tongue base), repeated on both sides.

   2.2- Efficacy of a lactoferrin mouthwash to attenuate the sensation of MT. Omur-Ozbeck et al. showed that a lactoferrin mouthwash completely attenuated an artificially-created MT by an iron sulphate mouthwash. For the investigator's patients, in case of spontaneous presence of a MT or after having artificially created it by the iron sulphate mouthwash, a lactoferrin mouthwash will be proposed and its efficacy to attenuate the MT will be evaluated.

   2.3- Psychophysical olfaction tests (European Test of olfactory Capacities ETOC from Thomas-Danguin T et al. Rhinology 2003;41:142-51) This test is constructed from odours contained in vials. It is made up of 16 series of 4 vials. In a series, only one of the four vials contains an odour. The patients must first find the vial which, among 4 contains the odour (test of detection) then in the vial chosen identify the odour (test of identification) among 4 alternatives proposed in the form of 4 verbal labels.
3. Impedancemetry Measurements of the spontaneous presence of a current in the oral cavity and the resistivity of the oral mucosa will be carried out by application of an electrode on the back of the tongue. This procedure is painless.
4. Evaluation of food intake by patients weighing, an analogic visual scale and of food pleasantness by MT specific questionnaire.
5. Characterization of quality of life through general EORTC QLQ30 and HNC-specific EORTC HNC35 quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Any head and neck cancer
* Before any treatment and treatment (surgery, chemotherapy, radiation therapy)
* Before the appearance of the metallic taste symptom
* Age ≥ 18 years
* Estimated life expectancy ≥ 6 months.
* Affiliation to a Social security system
* Patient who has given written consent signed before any specific procedure of the protocol

Exclusion Criteria:

* History of cancer (head and neck or other) that could be a confounding factor (dysgeusia, dysosmia, salivary composition disorder)
* Pregnant woman (frequent dysgeusia and dysosmia)
* Total laryngectomy (treatment-induced hyposmia)
* Early cancer recurrence (< 6 months after the end of the last treatment) because the taste, smell, and/or composition of the saliva can be altered by the cancer itself
* Persons deprived of liberty, under guardianship or under curatorship or unable to submit to the medical follow-up of the test for geographical, social or psychic reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with head and neck cancer before any treatment will be recruited. Repartition between the two groups will be performed a posteriori after onset or not of the metallic taste perception.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline salivary malondialdehyde level within one year after treatment completion | Day 0 (before any treatment), before the irradiation (about 1 month ½ after Day 0), half of the irradiation (approximately 3 months after Day 0), end of irradiation (approximately 4 months after Day 0), 6-10-14 and 16 months after Day 0
  The lipoperoxidation will be measured with salivary dosage of malondialdehyde (µmol/L). As metallic taste may vary according time, the measure will be repeated.

SECONDARY OUTCOMES:
Change from Baseline métabolites levels modifications of the saliva within one year after treatment completion | Day 0 (before any treatment), before the irradiation (about 1 month ½ after Day 0), half of the irradiation (approximately 3 months after Day 0), end of irradiation (approximately 4 months after Day 0), 6-10-14 and 16 months after Day 0
  Additional chemical modifications of the saliva will be tested by salivary dosages: uric acid in µmol/ml
Change from Baseline ions levels modifications of the saliva within one year after treatment completion | Day 0 (before any treatment), before the irradiation (about 1 month ½ after Day 0), half of the irradiation (approximately 3 months after Day 0), end of irradiation (approximately 4 months after Day 0), 6-10-14 and 16 months after Day 0
  Additional chemical modifications of the saliva will be tested by salivary dosages: Mn2+ and Zn2+, in µmol/ml
Change from Baseline enzymes levels modifications of the saliva within one year after treatment completion | Day 0 (before any treatment), before the irradiation (about 1 month ½ after Day 0), half of the irradiation (approximately 3 months after Day 0), end of irradiation (approximately 4 months after Day 0), 6-10-14 and 16 months after Day 0
  Additional chemical modifications of the saliva will be tested by salivary dosages: peroxydase, catalase, superoxide dismutase (in IU/ml)
Change from Baseline fungiform papillae density of the tonguewithin one year after treatment completion | Day 0 (before any treatment), before the irradiation (about 1 month ½ after Day 0), half of the irradiation (approximately 3 months after Day 0), end of irradiation (approximately 4 months after Day 0), 6-10-14 and 16 months after Day 0
  fungiform papillae density before, during and after treatment will be measured by tongue dermatoscopy. As metallic taste may vary according time, the measure will be repeated.
release of inhibition of the facial nerve on the glossopharyngeal nerve | Day 0 (before any treatment), before the irradiation (about 1 month ½ after Day 0), half of the irradiation (approximately 3 months after Day 0), end of irradiation (approximately 4 months after Day 0), 6-10-14 and 16 months after Day 0
  The release of inhibition of the facial nerve on the glossopharyngeal nerve will be tested with taste and smell psychophysical tests (supraliminory intensity taste testing and European Tests of Olfactory Capabilities) and a metallic taste-specific questionnaire [IJpma et al. Metallic Taste in Cancer Patients Treated with Systemic Therapy: A Questionnaire-based Study. Cancer Nutr 2017]. As metallic taste may vary according time, the measure will be repeated.
change from Baseline intraoral electric current within one year after treatment completion | Day 0 (before any treatment), before the irradiation (about 1 month ½ after Day 0), half of the irradiation (approximately 3 months after Day 0), end of irradiation (approximately 4 months after Day 0), 6-10-14 and 16 months after Day 0
  the presence of an intraoral electric current will be tested by impedancemetry. As metallic taste may vary according time, the measure will be repeated.
Change frome Baseline quality of life within one year after treatment completion | Day 0 (before any treatment), before the irradiation (about 1 month ½ after Day 0), half of the irradiation (approximately 3 months after Day 0), end of irradiation (approximately 4 months after Day 0), 6-10-14 and 16 months after Day 0
  questionnaires (EORTC QLQ30 and HN35). As quality of life may vary according time, the measure will be repeated.
Change frome Baseline food pleasantness and acceptability within one year after treatment completion | Day 0 (before any treatment), before the irradiation (about 1 month ½ after Day 0), half of the irradiation (approximately 3 months after Day 0), end of irradiation (approximately 4 months after Day 0), 6-10-14 and 16 months after Day 0
  questionnaires (IJpma el al. Nutrition and cancer. 2017;69:140-5) and an analogic visual scale of dietary intakes (from 1 to 10, from Thibault R et al. Clin Nutr. 2009;28:134-40). As metallic taste may vary according time, the measure will be repeated.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Feron, PhD, Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- CH Valence, Valence, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buiret G, Brignot H, Septier C, Thomas-Danguin T, Feron G. The nutritional impact of metallic taste in head and neck cancer patients: explorations and clinical implications. Support Care Cancer. 2024 Sep 11;32(10):651. doi: 10.1007/s00520-024-08854-z. PMID 39256281